CLINICAL TRIAL: NCT04519710
Title: Pilot, Interventional Study of the Specific Anti-HBV Vaccine Response After Vaccination in Patients Requiring Anti-CD20 Monoclonal Antibodies
Brief Title: Specific Anti-HBV Vaccine Response After Vaccination in Patients Requiring Anti-CD20 Monoclonal Antibodies
Acronym: HepB20
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Recherches et d'Etude sur la Pathologie Tropicale et le Sida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CREPATS 009
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: HBV
MeSH Terms: interventions — Rituximab; ocrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- multiple sclerosis or other inflammatory neurological disease (Experimental): HBV negative
  Interventions: Biological: o receive treatment with anti-CD20 (rituximab or ocrelizumab) and to be vaccinated against hepatitis B
- systemic vasculitis (Experimental): HBV negative
  Interventions: Biological: o receive treatment with anti-CD20 (rituximab or ocrelizumab) and to be vaccinated against hepatitis B
- an autoimmune disease (Experimental): HBV negative
  Interventions: Biological: o receive treatment with anti-CD20 (rituximab or ocrelizumab) and to be vaccinated against hepatitis B

INTERVENTIONS:
Biological: o receive treatment with anti-CD20 (rituximab or ocrelizumab) and to be vaccinated against hepatitis B — to receive treatment with anti-CD20 (rituximab or ocrelizumab) and to be vaccinated against hepatitis B

SUMMARY:
Vaccination coverage against HBV in France is around 30% in the adult population. Treatment with anti-CD20 is associated with a risk of reactivation of hepatitis B or acute or fulminant hepatitis in first-infected patients. HBV vaccination is recommended as before any anti-CD20 treatment in unimmunized patients.

However, there is no recommendation on which vaccination regimen to choose in patients on immunosuppressants / corticosteroids or with inflammatory or autoimmune disease.

For patients who have a need for rapid immunosuppressive therapy, the use of a standard vaccination schedule (D0, M1, M6) would be responsible for a loss of chance vis-à-vis the underlying disease with a delay of more than 6 months to start treatment with anti-CD20. An accelerated regimen (D0, D7, D21 and M12) allows healthy adults to obtain very rapid vaccine protection between 77 and 90.8%. The accelerated regimen can also be considered on a case-by-case basis in those adults with neurological pathologies, systemic vasculitis or autoimmune disease and who need to receive anti-CD20 antibodies if the combination of injections over a short period is likely to promote immunization.

The advantage of the accelerated regimen is to obtain 4 weeks, after the third dose of vaccine, anti-HBs antibodies at a protective level (> 10 IU / L) in approximately 77 to 90.8% of patients and in the general population. The booster injection at 12 months is essential for long-term protection.

DETAILED DESCRIPTION:
An accelerated regimen allows healthy adults to obtain vaccine protection very quickly. The accelerated regimen can also be considered on a case-by-case basis in those adults with neurological pathologies, systemic vasculitis or autoimmune disease requiring an anti-CD20 monoclonal antibody if the combination of injections over a short period is likely to promote immunization.

The aim of this pilot, interventional study is to evaluate the anti-HBV vaccine response measured by the level of anti-HBs antibodies greater than 10 IU / l after vaccination in patients to receive treatment with anti-CD20.

Evaluation of the specific anti-HBV vaccine response, measured by the level of anti-HBs antibodies greater than 10 IU / l at M2, M6 and M13 in patients having received a regimen accelerated by Engerix B 20 µg (D0, D7, J21), then recall 12 months later. Anti-CD20 drugs should be started at least 1 month after the first 3 injections for neurological pathologies and after the first 2 injections for vasculitis and autoimmune diseases (scheme linked to the underlying pathology with the need for rapid treatment with anti -CD20 in these pathologies).

Follow-up of 3 parallel cohorts of patients seronegative for hepatitis B virus (HBV):

* 1 cohort followed for multiple sclerosis or another inflammatory neurological disease (group 1)
* the cohort followed for systemic vasculitis (group 2)
* 1 cohort followed for an autoimmune disease (RA, Lupus, etc.) (group 3) to receive treatment with anti-CD20 (rituximab or ocrelizumab) and to be vaccinated against hepatitis B.

The patients will be followed for a period of 13 months after the start of the vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Multiple sclerosis or other known neurological disease (group 1), systemic vasculitis (group 2) or autoimmune disease (group 3)
* Decision on treatment with anti-CD20 (rituximab or ocrelizumab)
* Free and informed consent, oral
* Negative hepatitis B serology.

Exclusion Criteria:

* Previous hepatitis B vaccination
* Major disability
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Measure of the specific anti-HBV vaccine response, assessed by the level of anti-HBs antibodies greater than 10 IU / l at M2, M6 and M13 | 13 months
  regimen accelerated by Engerix B 20 µg (D0, D7, D21), then recall 12 months later
  regimen accelerated by Engerix B 20 µg (D0, D7, D21), then recall 12 months later regimen accelerated by HBV vaccine 20 µg (D0, D7, D21), then recall 12 months later

CONTACTS AND LOCATIONS:
Overall Officials: valérie Pourcher, MD, Principal Investigator — Pitie-Salpetriere Hospital
Locations (1):
- Valérie POURCHER, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No